CLINICAL TRIAL: NCT00513305
Title: An Open-Label, Randomized Study of Low-Dose Cytarabine in Combination With Arsenic Trioxide Compared With Low-Dose Cytarabine Alone for the Treatment of Elderly Patients With Acute Myeloid Leukemia
Brief Title: Cytarabine in Combination With Arsenic Trioxide vs. Cytarabine Alone in Elderly Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has been stopped by sponsor decision
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C18477/3059/AM/US-CA
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia, cytarabine, arsenic trioxide.
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Arsenic Trioxide; Cytarabine

ARMS (2):
- Low-dose cytarabine plus arsenic trioxide (Active Comparator): Cycle 1 cytarabine 10 mg/m^2 was administered subcutaneously (sc) twice daily (bid) on days 1-14. 0.25 mg/kg arsenic trioxide was administered intravenously (iv) on days 1-5 and days 8-12. Cycle 2 A second identical cycle of cytarabine and arsenic trioxide was given to patients with persistent disease. Patients who achieved complete remission (CR), complete remission with incomplete platelet count recovery (CRp), or partial remission (PR) after 1 or 2 cycles received a 14-day consolidation cycle of cytarabine and arsenic trioxide with the doses and schedule identical to the initial cycle. A recovery period of up to 4 weeks between the attainment of CR, CRp, or PR and the initiation of consolidation treatment was allowed. Patients who completed consolidation treatment started maintenance treatment of arsenic trioxide 0.25 mg/kg iv on days 1 and 4 and cytarabine 10 mg/m^2 sc bid on days 1 through 7 of a 28-day cycle.
  Interventions: Drug: Arsenic trioxide; Drug: Low-dose cytarabine alone
- Low-dose cytarabine alone (Active Comparator): Cytarabine was administered at a dose of 10 mg/m^2 sc bid from days 1-14 of cycle 1. A second identical cycle of cytarabine was given to patients with persistent disease. Patients who achieved a complete remission (CR), complete remission with incomplete platelet count recovery (CRp), or partial remission (PR) after 1 or 2 cycles received a 14-day consolidation cycle of cytarabine with the doses and schedule identical to the initial treatment cycle. Recovery period up to 4 weeks between the attainment of CR, CRp, or PR and the initiation of consolidation treatment was allowed. Patients who completed consolidation treatment started maintenance treatment of cytarabine at 10 mg/m^2 sc bid on days 1-7 of a 28-day cycle. Patients started maintenance treatment within 42 days after platelet count recovery. Maintenance treatment continued for 2 years or until unacceptable toxicity or disease progression.
  Interventions: Drug: Low-dose cytarabine alone

INTERVENTIONS:
Drug: Arsenic trioxide — Arsenic trioxide will be administered intravenously (iv) at a dose of 0.25 mg/kg.
  Arms: Low-dose cytarabine plus arsenic trioxide
Drug: Low-dose cytarabine alone — Cytarabine will be administered at a dose of 10 mg/m^2 subcutaneously (sc) twice a day (bid).

SUMMARY:
The primary objective of this study is to determine whether low-dose cytarabine in combination with arsenic trioxide is more effective than low-dose cytarabine alone in achieving complete remission in elderly patients (≥60 years of age) with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* The patient has confirmed acute myeloid leukemia (AML).
* The patient is unwilling or unable to tolerate conventional induction chemotherapy.
* The patient has no comorbid conditions that would limit life expectancy to less than 3 months.
* Patient must meet specific laboratory parameters for study inclusion.

Exclusion Criteria:

- The patient has had previous cytotoxic chemotherapy for acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

Previous treatment with low-dose cytarabine is not permitted.

* The patient has a QT interval outside of the protocol-specified range.
* The patient has laboratory values outside of protocol-specified ranges.
* The patient is concurrently treated with cytotoxic therapy, radiation, or investigational agents.
* The patient has uncontrolled, severe cardiovascular or pulmonary disease or other uncontrolled medical condition.
* The patient has known central nervous system involvement with AML.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - USC / Norris Cancer Hospital, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of Illinois, Chicago, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Brody School of Medicine, Greenville, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Health Science Center, San Antonio, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven centers in the United States and one center in Canada. First patient enrolled 12 October 2007; last patient completed protocol-specified treatment 5 July 2009; last patient completed survival follow-up contact 16 December 2009.
Groups:
- Low-dose Cytarabine Plus Arsenic Trioxide: Cycle 1. 10 mg/m^2 cytarabine was administered subcutaneously (sc) twice daily (bid) on days 1-14. 0.25 mg/kg arsenic trioxide was administered intravenously (iv) on days 1-5 and days 8-12. Cycle 2. A second identical cycle of cytarabine and arsenic trioxide was given to patients with persistent disease identified from a bone marrow sample taken on day 21 of cycle 1. Patients who achieved complete remission (CR), complete remission with incomplete platelet count recovery (CRp), or partial remission (PR) after 1 or 2 cycles received a 14-day consolidation cycle of cytarabine and arsenic trioxide with the doses and schedule identical to the initial cycle. A recovery period of up to 4 weeks between the attainment of CR, CRp, or PR and the initiation of consolidation treatment was allowed. Patients who completed consolidation treatment started maintenance treatment of arsenic trioxide 0.25 mg/kg iv on days 1 and 4 and cytarabine 10 mg/m^2 sc bid on days 1 through 7 of a 28-day cycle.
- Low-dose Cytarabine Alone: Cytarabine was administered at a dose of 10 mg/m^2 sc bid from days 1-14 of cycle 1. A second identical cycle of cytarabine treatment was given to patients with persistent disease identified from a bone marrow sample taken on day 21 of cycle 1. Patients who achieved a complete remission (CR), complete remission with incomplete platelet count recovery (CRp), or partial remission (PR) after 1 or 2 cycles received a 14-day consolidation cycle of cytarabine with the doses and schedule identical to the initial treatment cycle. A recovery period of up to 4 weeks between the attainment of CR, CRp, or PR and the initiation of consolidation treatment was allowed. Patients who completed consolidation treatment started maintenance treatment of cytarabine at 10 mg/m^2 sc bid on days 1-7 of a 28-day cycle. Patients started maintenance treatment within 42 days after platelet count recovery. Maintenance treatment continued for 2 years or until unacceptable toxicity or disease progression.
Period: Overall Study
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Started | 33 | 34 (One subject withdrew prior to receiving study medication)
Completed | 5 | 7
Not Completed | 28 | 27
Not completed — Adverse Event | 6 | 2
Not completed — Death (through Consolidation Treatment) | 2 | 2
Not completed — Lack of Efficacy | 8 | 13
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease progression | 8 | 5
Not completed — Eligible for stem cell transplant | 1 | 0
Not completed — Hematologic counts did not recover | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Persistent hypocellularity | 0 | 1
Not completed — Sponsor Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 24 | 27 | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 70.9 (7.1) | 71.5 (6.8) | 71.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64
  Canada | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Complete Remission (CR)
Description: The primary efficacy variable was the percentage of subjects in each treatment group who achieved complete remission after treatment with study drug. Complete remission was defined as: 1) Less than 5% blasts in normocellular bone marrow sample. 2) No blasts in bone marrow sample containing Auer rods. 3)Clearance of previous extramedullary disease. 4)Normal values for absolute neutrophil count (at least 1000/microliter), platelet count (at least 100,000/microliter), without platelet transfusions, and in absence of peripheral myeloblasts.
Time Frame: From baseline through Day 70. Assessments were performed on Day 21 in cycle 1, no later than Day 56 of cycle 1 or 2 (if applicable), and no later than Day 70 of cycle 1 or 2 (if applicable) or at any other time at the discretion of the investigator
Population: Intention to treat (ITT) Analysis Set
Measure: Number; unit: Percentage of participants in CR
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Number analyzed (Participants) | 33 | 34
Percentage of participants in CR | 15.2 [0.051 to 0.319] | 8.8 [0.019 to 0.0237]
Statistical Analysis 1: Comparison: Low-dose Cytarabine Plus Arsenic Trioxide vs Low-dose Cytarabine Alone; The hypothesis of equal complete remission rates between the two treatment groups was tested using a 2-sided, normal approximation to the difference in binomial proportions test with two-sided alpha equal to 0.05; Test type: Superiority or Other; p = 0.425, Chi-squared — The p-value is from the Pearson chi-square test for testing the equality of two binomial proportions, assuming normal approximation of the binomial proportions; There were no adjustments for covariates. Since the primary endpoint was prespecified, no adjustment for multiplicity of endpoints was introduced

2. Secondary Outcome: Number of Participants Who Died or Were Censored by 24 Months
Description: This measure (time to death or censor) was defined for all enrolled subjects from the date of randomization until death from any cause. If a subject was not known to have died by the end of the followup period, observation of overall survival was censored on the date the patient was last known to be alive. The number of participants who died or were censored is presented here. (Note: all subjects participating in this study had either died or were censored by 24 months.)
Time Frame: From Baseline through 24 months following Baseline
Measure: Number; unit: Participants
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Number analyzed (Participants) | 33 | 34
Participants | 33 | 34
Statistical Analysis 1: Comparison: Low-dose Cytarabine Plus Arsenic Trioxide vs Low-dose Cytarabine Alone; Test type: Superiority or Other; p = 0.829, Log Rank; Cox Proportional Hazard = 1.027, 95% CI 2-sided [0.535 to 1.973]

3. Secondary Outcome: Proportion of Participants With Relapse-Free Survival (RFS)Using the Kaplan-Meier Estimate
Description: RFS is defined for patients who achieved a complete remission (CR), complete remission with incomplete platelet recovery (CRp), or partial remission(PR), and was measured from the date of attaining CR, CRp, or PR until the date of AML relapse or death from any cause, whichever occurred first. For a patient not known to have relapsed or died by the end of the study followup, observation of relapse free survival was censored on the date of the last followup examination. The Kaplan Meier Estimate of relapse-free survival at Month 3 and Month 6 is presented here.
Time Frame: From Baseline (randomization) through 24 months following Baseline
Population: Population analyzed are the subjects who who achieved a complete remission (CR), complete remission with incomplete platelet recovery (CRp), or partial remission(PR)during the course of the study
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Number analyzed (Participants) | 21 | 29
Proportion of participants
  Month 3 (95% Confidence Interval) | 0.818 [0.447 to 0.951] | 0.800 [0.204 to 0.969]
  Month 6 (95% Confidence Interval) | 0.818 [0.447 to 0.951] | 0.800 [0.204 to 0.969]
Statistical Analysis 1: Comparison: Low-dose Cytarabine Plus Arsenic Trioxide vs Low-dose Cytarabine Alone; Test type: Superiority or Other; p = 0.527, Log Rank; Cox Proportional Hazard = 2.310, 95% CI 2-sided [0.160 to 33.343] — Estimate based on Cox Proportional Hazards Model adjusting for age, Eastern Cooperative Oncology Group (ECOG) status, white blood count and presence of antecedent hematologic disorder

4. Secondary Outcome: Number of Participants Who Experienced Early Death
Description: Early death is defined as death from any cause within the first 14 days after start of study drug treatment. The number of patients in each study group who experienced early death is presented here.
Time Frame: 14 days from start of study drug treatment
Measure: Number; unit: Participants
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Number analyzed (Participants) | 33 | 34
Participants | 0 | 2

5. Secondary Outcome: Number of Participants Who Experienced Induction (Thirty-Day) Mortality
Description: The number of subjects who died from any cause within the first 30 days after the start of study drug treatment is presented here.
Time Frame: Up to 30 days following start of study drug treatment
Measure: Number; unit: Participants
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Number analyzed (Participants) | 33 | 34
Participants | 3 | 2

6. Secondary Outcome: Proportion of Participants Surviving at 6 Months and 12 Months Using the Kaplan Meier Estimate
Description: The duration of overall survival was defined for all patients and was measured from the date of randomization until death from any cause. For a patient who was not known to have died by the end of the follow-up period, observation of overall survival was censored on the date the patient was last known to be alive. The estimate of likelihood of survival at 6 and 12 months after Baseline using the Kaplan Meier Estimate is presented here.
Time Frame: Baseline through 12 months
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Number analyzed (Participants) | 33 | 34
Proportion of Participants
  Month 6 (95% Confidence Interval) | 0.626 [0.435 to 0.768] | 0.649 [0.454 to 0.789]
  Month 12 (95% Confidence Interval) | 12.22 [4.37 to 16.76] | 8.51 [5.72 to 19.65]
Statistical Analysis 1: Comparison: Low-dose Cytarabine Plus Arsenic Trioxide vs Low-dose Cytarabine Alone; Test type: Superiority or Other; p = 0.8289, Log Rank; Cox Proportional Hazard = 1.027, 95% CI 2-sided [0.535 to 1.973] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: approximately 2 years
Description: Adverse events were collected from the date the ICF was signed through 30 days after the last dose of study drug.
Arm/Group | Low-dose Cytarabine Plus Arsenic Trioxide | Low-dose Cytarabine Alone
Serious Adverse Events (participants affected / at risk) | 19/33 | 21/33
Other Adverse Events (participants affected / at risk) | 33/33 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Cytarabine Plus Arsenic Trioxide (N=33) | Low-dose Cytarabine Alone (N=33)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abscess bacterial (Infections and infestations) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 9 (9)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia fungal (Infections and infestations) | 2 (2) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Cytarabine Plus Arsenic Trioxide (N=33) | Low-dose Cytarabine Alone (N=33)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Asthenia (General disorders) | 7 (7) | 9 (9)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Bacteraemia (Infections and infestations) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 2 (2)
Blood culture positive (Investigations) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Breath sounds abnormal (Investigations) | 3 (3) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac murmur (Investigations) | 1 (1) | 2 (2)
Catheter site erythema (General disorders) | 4 (4) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Chest pain (General disorders) | 5 (5) | 6 (6)
Chills (General disorders) | 5 (5) | 7 (7)
Clostridial infection (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 14 (14) | 11 (11)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 21 (21) | 14 (14)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4)
Dysarthria (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Enterococcal infection (Infections and infestations) | 0 (0) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fatigue (General disorders) | 10 (10) | 9 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 16 (16)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 3 (3) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 10 (10) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1)
Liver function test abnormal (Investigations) | 5 (5) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Mucosal inflammation (General disorders) | 4 (4) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (15) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oedema (General disorders) | 6 (6) | 0 (0)
Oedema peripheral (General disorders) | 16 (16) | 14 (14)
Oral candidiasis (Infections and infestations) | 2 (2) | 2 (2)
Pain (General disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 9 (9) | 12 (12)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 6 (6) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 7 (7)
Weight decreased (Investigations) | 4 (4) | 4 (4)
Weight increased (Investigations) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3)
Confusional state (Psychiatric disorders) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 5 (5)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Oliguria (Renal and urinary disorders) | 0 (0) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Rales (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 10 (10) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Blood blister (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 13 (13) | 9 (9)
Haematoma (Vascular disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
In September 2009, the sponsor decided to stop the study due to difficulty in enrollment. The study was stopped prior to the first planned interim analysis. Most of the analysis planned in the protocol was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days